CLINICAL TRIAL: NCT03027037
Title: Perinatal Emotion and Relationships Longitudinal Study
Acronym: PEARLS
Status: Completed | Type: Observational
Sponsor: University of Colorado, Boulder (Other)
Collaborators: John Templeton Foundation (Other); Emory University (Other); University of Michigan (Other); Columbia University (Other); Queen's University (Other)
Responsible Party: Principal Investigator, Sona Dimidjian, Professor and Director, University of Colorado, Boulder
Other Study IDs: 49683
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Remitted Major Depression Group: Women in this group will have experienced at least one episode of major depression in their lifetime, but no episodes in the two months prior to study enrollment.
- Control Group: Women in this group will never have experienced any Diagnostic and Statistical Manual of Mental Disorders, 5th Edition Axis I psychological disorder.

SUMMARY:
This study, funded by the John Templeton Foundation, will examine birth and the early postpartum period (BEPP) as a transformative life experience that may shift women's experience of emotion in such ways as to a) support enhanced other-oriented emotions and b) underlie risk or resilience from psychopathology.

DETAILED DESCRIPTION:
Specifically, the study will investigate the extent to which women can accurately have knowledge about and predict changes in self- and other-oriented emotion processes associated with BEPP. The investigators will also characterize the extent to which BEPP changes self- and other-oriented emotion processes and self- and other-oriented social behaviors. Further, the investigators will identify distinct trajectories of change in cognitive processes and self- and other-oriented emotion processes related to BEPP, and examine how those trajectories are associated with psychological adjustment (e.g., risk and relapse of psychopathology). Finally, the investigators will identify which particular features of BEPP are related to distinct patterns of change in self- and other-oriented emotion processes.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Female
* Currently pregnant - approximately no more than 34 weeks gestational age
* Able to read and write in English fluently
* MDD Group: Meet DSM-IV/DSM-5 criteria for at least 1 past episode of Major Depressive Disorder
* MDD Group: DO NOT meet DSM-IV/DSM-5 criteria for any episodes of Major Depressive Disorder in past 2 months (currently in symptom remission)

Exclusion Criteria:

* Previous birth to a living child (i.e., this pregnancy is not their first child)
* Imminently suicidal or homicidal
* History of severe head trauma, stroke, neurological disease
* History of brain tumors or surgery
* Severe medical illness (e.g., autoimmune disorder, blindness, cardiovascular disease, HIV/AIDS)
* Endocrine disorders (e.g., Cushing's disease, thyroid disorder)
* Alcohol/substance abuse or dependence within the past six months
* Current psychotic episode (impairing ability to consent, participate, or keep patient and experimenter safe)
* Inability to follow study procedures
* CTL Group: Current or lifetime Axis I disorder (i.e., anxiety disorders, major depression, mania/hypomania, dysthymia, schizophrenia, schizoaffective disorder, substance abuse/dependence, eating disorders, hypochondriasis, pain disorder, or adjustment disorders)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include up to 200 pregnant adult women over the age of 18 across the United States. Two roughly equal groups of participants will be recruited: women with a history of major depressive disorder, currently in remission (MDD) and healthy controls with no current or lifetime history of mental illness (CTL).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of mood episodes and anxiety disorders | Throughout study (pregnancy to 6 months postpartum)
  Assessed via interview
Mood and anxiety symptoms | Throughout study (pregnancy to 6 months postpartum)
  Assessed via questionnaires
Emotion reactivity and regulation | Throughout study (pregnancy to 6 months postpartum)
  Assessed via questionnaires, experimental tasks, and physiological measurement
Empathic accuracy | Throughout study (pregnancy to 6 months postpartum)
  Assessed via experimental tasks
Prosocial behavior | Throughout study (pregnancy to 6 months postpartum)
  Assessed via questionnaires and experimental tasks
Well-being and social support | Throughout study (pregnancy to 6 months postpartum)
  Assessed via questionnaires
Parenting sensitivity, efficacy, stress, bond with infant | Throughout study (pregnancy to 6 months postpartum)
  Assessed via questionnaires and behavioral observation

CONTACTS AND LOCATIONS:
Overall Officials: Sona Dimidjian, PhD, Principal Investigator — University of Colorado, Boulder; June Gruber, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No